CLINICAL TRIAL: NCT03067844
Title: Effects of the PCSK9 Antibody AliroCuMab on Coronary Atherosclerosis in PatieNts With Acute Myocardial Infarction: A Serial, Multivessel, Intravascular Ultrasound, Near-Infrared Spectroscopy And Optical Coherence Tomography Imaging Study
Brief Title: Vascular Effects of Alirocumab in Acute MI-Patients
Acronym: PACMAN-AMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-01382
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Coronary Vessel; Coronary Circulation; Atheroma; Myocardial
MeSH Terms: conditions — Plaque, Atherosclerotic | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alirocumab (Experimental): Alirocumab 150 mg/mL, pre-filled auto-injector pen, every second week, starting at day 1 and up to week 50.
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): Placebo, pre-filled auto-injector pen, every second week, starting at day 1 and up to week 50.
  Interventions: Drug: Alirocumab

INTERVENTIONS:
Drug: Alirocumab — Pre-filled auto-injector pen every second week, starting at day 1 and up to week 50

SUMMARY:
Coronary artery disease (CAD) is the most frequent cause of mortality in the industrialized world. Hypercholesterolemia is a major risk factor for the development and progression of CAD. While statins currently represent the first-line, gold-standard therapy for primary and secondary prevention of cardiovascular morbidity and mortality, nearly 50% of patients in Europe and Canada treated with statins do not achieve their target levels of low-density lipoprotein cholesterol (LDL-C) or cannot tolerate effective statin doses.

Recently, a growing number of studies of PCSK9 inhibitors in a wide spectrum of patients with hyperlipidemia on or off lipid-lowering therapy, familial hypercholesterolemia, and statin intolerance demonstrated consistent, profound, and sustained reductions in LDL-C with greater magnitude of reduction as compared with high-dose statin regimens. However, the effects of PCSK9 inhibition on coronary plaque morphology remain unknown.

This study will investigate the effect of the PCSK9 inhibitor alirocumab in patients with acute myocardial infarction undergoing percutaneous coronary intervention (PCI) in the infarct-related artery and receiving guideline-recommended high-intensity statin therapy. A serial, multivessel, intravascular ultrasound, near-infrared spectroscopy and optical coherence tomography imaging study will be performed to determine the change in plaque volume at week 52. A total of 294 patients will be enrolled in the study and randomized in a 1:1 ratio to either alirocumab or placebo.

DETAILED DESCRIPTION:
Substudies

* Biobank/drug monitoring, all sites
* Lipidomics (n=294), all sites
* Platelet Function (n=~150), Bern
* Endothelial Function (n=~150), Bern
* Neatherosclerosis (n=~294), all sites
* Neutrophilic Extracellular Trap (NET), (n=~50), Vienna
* OCT-NIRS/IVUS Matching Substudy (n=~104), Bern
* Positron Emission Computed Tomography (PET-CT), (n=~50), Copenhagen
* Shear Stress (n=~294), London
* Quantitative Flow Ratio (QFR) (n=~294), Bern

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years at screening;
* Acute myocardial infarction: acute ST-segment elevation myocardial infarction (STEMI) with pain onset within ≤24h, or non-ST segment elevation myocardial infarction (NSTEMI), with at least one coronary segment (culprit lesion) requiring PCI;
* LDL-C ≥70 mg/dL (≥1.8 mmol/L) assessed prior to, or during PCI in patients who have been receiving any stable statin regimen within ≥ 4 weeks prior to enrollment; OR LDL-C ≥125 mg/dL (≥3.2 mmol/L) in patients who are statin-naïve or have not been on stable statin regimen for ≥ 4 weeks prior to enrollment;
* At least two major native coronary arteries ("target vessels") each meeting the following criteria for intracoronary imaging immediately following the qualifying PCI procedure: Angiographic evidence of <50% reduction in lumen diameter by angiographic visual estimation;
* Target vessel deemed to be accessible to imaging catheters and suitable for intracoronary imaging in the proximal (50mm) segment ("target segment");
* Target vessel may not be a bypass (saphenous vein or arterial) graft or a bypassed native vessel;
* Target vessel must not have undergone previous PCI within the target segment;
* Target vessel is not candidate for intervention at the time of qualifying PCI or over the following 6 months in the judgment of the Investigator;
* Hemodynamic stability allowing the repetitive administration of nitroglycerine;
* Ability to understand the requirements of the study and to provide informed consent;
* Willingness to undergo follow-up intracoronary imaging.

Exclusion Criteria:

* Left-main disease, defined as ≥50% reduction in lumen diameter of the left main coronary artery by angiographic visual estimation;
* Three-vessel disease, defined as ≥70% reduction in lumen diameter of three major epicardial coronary arteries by angiographic visual estimation or in major branches of one or more of these arteries, irrespective of the localization (proximal 50mm or more distal localization) of the obstructive lesions;
* History of coronary artery bypass surgery;
* "Thrombolysis In Myocardial Infarction" (TIMI) flow <2 of the infarct-related artery after PCI;
* Unstable clinical status (hemodynamic or electrical instability);
* Significant coronary calcification or tortuosity deemed to preclude IVUS, NIRS and OCT evaluation;
* Uncontrolled cardiac arrhythmia, defined as recurrent and symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response not controlled by medications in the past 3 months prior to screening;
* Severe renal dysfunction, defined by estimated glomerular filtration rate <30 ml/min/1.73m2;
* Active liver disease or hepatic dysfunction;
* Known intolerance to rosuvastatin OR known statin intolerance;
* Known allergy to contrast medium, heparin, aspirin, ticagrelor or prasugrel;
* Known sensitivity to any substances to be administered, including known statin intolerance;
* Patients who previously received alirocumab or other PCSK9 inhibitor;
* Patient who received cholesterol ester transfer protein inhibitors in the past 12 months prior to screening;
* Treatment with systemic steroids or systemic cyclosporine in the past 3 months;
* Known active infection or major hematologic, metabolic, or endocrine dysfunction in the judgment of the Investigator;
* Planned surgery within 12 months;
* Patients who will not be available for study-required visits in the judgment of the Investigator;
* Current enrollment in another investigational device or drug study;
* History of cancer within the past 5 years, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer;
* Estimated life expectancy less than 1 year;
* Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Change in percent atheroma volume (PAV) | Baseline to week 52
  Change in PAV by greyscale intravascular ultrasound (IVUS)

SECONDARY OUTCOMES:
Change in total lipid-core burden index (LCBItotal) | Baseline to week 52
  Change in LCBItotal as determined by near infrared spectroscopy (NIRS)
Change in maximum LCBI in any 4-mm segment (Powered) | Baseline to week 52
  Change in maximum LCBI in any 4-mm segment (maxLCBI4mm) as determined by NIRS
Change in minimal fibrous cap thickness (Powered) | Baseline to week 52
  Change in minimal fibrous cap thickness as determined by optical coherence tomography (OCT)
Change in mean fibrous cap thickness | Baseline to week 52
  Change in mean fibrous cap thickness as determined by OCT
Change in average angular extension (AAE) of macrophages | Baseline to week 52
  Change in AAE of macrophages as determined by OCT
Change in normalized total atheroma volume (NTAV) | Baseline to week 52
  Change in NTAV by IVUS
Change in LDL-cholesterol | Baseline to week 52
  Change in LDL-cholesterol
Change in hsCRP | Baseline to week 52
  Change in hsCRP
Change in high sensitivity troponin T (hsTnT) | Baseline to week 52
  Change in hsTnT
Change in N-terminal prohormone of brain natriuretic peptide (NT-pro-BNP) | Baseline to week 52
  Change in NT-pro-BNP
Change in further biomarkers | Baseline to week 52
  Change in lipid and inflammatory markers and their association with indices of plaque progression/regression
Death | Baseline to week 52
  Any death, cardiac death
Non-fatal myocardial infarction | Baseline to week 52
  Any non-fatal myocardial infarction
Ischemia-driven coronary revascularization | Baseline to week 52
  Any ischemia-driven coronary revascularization
Stroke | Baseline to week 52
  Any ischemic stroke/transient ischemic attack

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Raeber, Prof., MD, Principal Investigator — Bern Universitiy Hospital
Locations (9):
- University Hospital Vienna (AKH), Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- Netherlands (2):
  - Radboud Univerity, Nijmegen Medical Centre, Nijmegen, Gelderland
  - Erasmus Thoraxcentre, Rotterdam
- Switzerland (5):
  - Basel University Hospital, Basel
  - Bern University Hospital Inselspital, Bern
  - Hopitaux Universitaires Geneve, Geneva
  - Stadtspital Triemli, Zurich
  - University Hospital Zurich USZ, Zurich

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJP, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Honda S, Shishikura D, Scherer DJ, Borgman M, Brennan DM, Wolski K, Nissen SE. Effect of Evolocumab on Coronary Plaque Composition. J Am Coll Cardiol. 2018 Oct 23;72(17):2012-2021. doi: 10.1016/j.jacc.2018.06.078. PMID 30336824
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Result] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923
- [Result] Cannon CP, Cariou B, Blom D, McKenney JM, Lorenzato C, Pordy R, Chaudhari U, Colhoun HM; ODYSSEY COMBO II Investigators. Efficacy and safety of alirocumab in high cardiovascular risk patients with inadequately controlled hypercholesterolaemia on maximally tolerated doses of statins: the ODYSSEY COMBO II randomized controlled trial. Eur Heart J. 2015 May 14;36(19):1186-94. doi: 10.1093/eurheartj/ehv028. Epub 2015 Feb 16. PMID 25687353
- [Result] Kastelein JJ, Ginsberg HN, Langslet G, Hovingh GK, Ceska R, Dufour R, Blom D, Civeira F, Krempf M, Lorenzato C, Zhao J, Pordy R, Baccara-Dinet MT, Gipe DA, Geiger MJ, Farnier M. ODYSSEY FH I and FH II: 78 week results with alirocumab treatment in 735 patients with heterozygous familial hypercholesterolaemia. Eur Heart J. 2015 Nov 14;36(43):2996-3003. doi: 10.1093/eurheartj/ehv370. Epub 2015 Sep 1. PMID 26330422
- [Result] Robinson JG, Farnier M, Krempf M, Bergeron J, Luc G, Averna M, Stroes ES, Langslet G, Raal FJ, El Shahawy M, Koren MJ, Lepor NE, Lorenzato C, Pordy R, Chaudhari U, Kastelein JJ; ODYSSEY LONG TERM Investigators. Efficacy and safety of alirocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1489-99. doi: 10.1056/NEJMoa1501031. Epub 2015 Mar 15. PMID 25773378
- [Result] Koskinas KC, Ughi GJ, Windecker S, Tearney GJ, Raber L. Intracoronary imaging of coronary atherosclerosis: validation for diagnosis, prognosis and treatment. Eur Heart J. 2016 Feb 7;37(6):524-35a-c. doi: 10.1093/eurheartj/ehv642. Epub 2015 Dec 11. PMID 26655874
- [Result] Raber L, Taniwaki M, Zaugg S, Kelbaek H, Roffi M, Holmvang L, Noble S, Pedrazzini G, Moschovitis A, Luscher TF, Matter CM, Serruys PW, Juni P, Garcia-Garcia HM, Windecker S; IBIS 4 (Integrated Biomarkers and Imaging Study-4) Trial Investigators (NCT00962416). Effect of high-intensity statin therapy on atherosclerosis in non-infarct-related coronary arteries (IBIS-4): a serial intravascular ultrasonography study. Eur Heart J. 2015 Feb 21;36(8):490-500. doi: 10.1093/eurheartj/ehu373. Epub 2014 Sep 2. PMID 25182248
- [Result] Pu J, Mintz GS, Brilakis ES, Banerjee S, Abdel-Karim AR, Maini B, Biro S, Lee JB, Stone GW, Weisz G, Maehara A. In vivo characterization of coronary plaques: novel findings from comparing greyscale and virtual histology intravascular ultrasound and near-infrared spectroscopy. Eur Heart J. 2012 Feb;33(3):372-83. doi: 10.1093/eurheartj/ehr387. Epub 2011 Oct 20. PMID 22019821
- [Result] Maehara A, Cristea E, Mintz GS, Lansky AJ, Dressler O, Biro S, Templin B, Virmani R, de Bruyne B, Serruys PW, Stone GW. Definitions and methodology for the grayscale and radiofrequency intravascular ultrasound and coronary angiographic analyses. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S1-9. doi: 10.1016/j.jcmg.2011.11.019. PMID 22421222
- [Result] Madder RD, Goldstein JA, Madden SP, Puri R, Wolski K, Hendricks M, Sum ST, Kini A, Sharma S, Rizik D, Brilakis ES, Shunk KA, Petersen J, Weisz G, Virmani R, Nicholls SJ, Maehara A, Mintz GS, Stone GW, Muller JE. Detection by near-infrared spectroscopy of large lipid core plaques at culprit sites in patients with acute ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2013 Aug;6(8):838-46. doi: 10.1016/j.jcin.2013.04.012. Epub 2013 Jul 17. PMID 23871513
- [Result] Raber L, Zanchin T, Baumgartner S, Taniwaki M, Kalesan B, Moschovitis A, Garcia-Garcia HM, Justiz J, Pilgrim T, Wenaweser P, Meier B, Juni P, Windecker S. Differential healing response attributed to culprit lesions of patients with acute coronary syndromes and stable coronary artery after implantation of drug-eluting stents: an optical coherence tomography study. Int J Cardiol. 2014 May 1;173(2):259-67. doi: 10.1016/j.ijcard.2014.02.036. Epub 2014 Feb 28. PMID 24631113
- [Result] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Derived] Schmidt LE, Burnap SA, Singh B, Takov K, Losdat S, Schrutka L, Galli L, Theofilatos K, Otto GW, Hengstenberg C, Tzoulaki I, Lang IM, Koskinas KC, Speidl WS, Raber L, Mayr M. Integrative Proteomic and Lipidomic Analysis of Post-Myocardial Infarction Patients Treated With PCSK9 Antibodies and Statins. Circ Genom Precis Med. 2026 Feb 10:e005345. doi: 10.1161/CIRCGEN.125.005345. Online ahead of print. PMID 41664920
- [Derived] van der Velpen V, Haner JD, Kakizaki R, Bar S, Ueki Y, Siontis GCM, Stortecky S, Biccire FG, Ambuhl M, Kaiser C, Iglesias JF, Mach F, van Geuns RJ, Daemen J, Engstrom T, Ondracek AS, Lang I, Bourantas CV, Matter CM, Windecker S, Koskinas KC, Mayr M, Losdat S, Raber L, Haschke M, Spirk D. Intake of high-intensity statin after acute myocardial infarction assessed by direct drug concentration measurement: association with LDL-C response and coronary plaque modifications in the PACMAN-AMI trial. Eur J Prev Cardiol. 2025 Aug 12:zwaf457. doi: 10.1093/eurjpc/zwaf457. Online ahead of print. PMID 40796144
- [Derived] Koskinas KC, Haner J, Ueki Y, Otsuka T, Lonborg J, Shibutani H, Kakizaki R, Kaiser C, van Geuns RJ, Ondracek AS, Praz F, Ambuhl M, Spirk D, Lanz J, Daemen J, Heg D, Mayr M, Mach F, Windecker S, Engstrom T, Lang IM, von Eckardstein A, Losdat S, Raber L. Association of Lipoprotein(a) With Changes in Coronary Atherosclerosis in Patients Treated With Alirocumab. Circ Cardiovasc Imaging. 2024 Nov;17(11):e016683. doi: 10.1161/CIRCIMAGING.124.016683. Epub 2024 Nov 19. PMID 39561225
- [Derived] Biccire FG, Kakizaki R, Koskinas KC, Ueki Y, Haner J, Shibutani H, Lonborg J, Spitzer E, Iglesias JF, Otsuka T, Siontis GCM, Stortecky S, Kaiser C, Ambuhl M, Morf L, Ondracek AS, van Geuns RJ, Spirk D, Daemen J, Mach F, Windecker S, Engstrom T, Lang I, Losdat S, Raber L. Lesion-Level Effects of LDL-C-Lowering Therapy in Patients With Acute Myocardial Infarction: A Post Hoc Analysis of the PACMAN-AMI Trial. JAMA Cardiol. 2024 Dec 1;9(12):1082-1092. doi: 10.1001/jamacardio.2024.3200. PMID 39221516
- [Derived] Rexhaj E, Bar S, Soria R, Ueki Y, Haner JD, Otsuka T, Kavaliauskaite R, Siontis GC, Stortecky S, Shibutani H, Spirk D, Engstrom T, Lang I, Morf L, Ambuhl M, Windecker S, Losdat S, Koskinas KC, Raber L; PACMAN-AMI Investigators. Effects of alirocumab on endothelial function and coronary atherosclerosis in myocardial infarction: A PACMAN-AMI randomized clinical trial substudy. Atherosclerosis. 2024 May;392:117504. doi: 10.1016/j.atherosclerosis.2024.117504. Epub 2024 Mar 6. PMID 38513436
- [Derived] Biccire FG, Haner J, Losdat S, Ueki Y, Shibutani H, Otsuka T, Kakizaki R, Hofbauer TM, van Geuns RJ, Stortecky S, Siontis GCM, Bar S, Lonborg J, Heg D, Kaiser C, Spirk D, Daemen J, Iglesias JF, Windecker S, Engstrom T, Lang I, Koskinas KC, Raber L. Concomitant Coronary Atheroma Regression and Stabilization in Response to Lipid-Lowering Therapy. J Am Coll Cardiol. 2023 Oct 31;82(18):1737-1747. doi: 10.1016/j.jacc.2023.08.019. Epub 2023 Aug 26. PMID 37640248
- [Derived] Bar S, Kavaliauskaite R, Otsuka T, Ueki Y, Haner JD, Siontis GCM, Stortecky S, Shibutani H, Temperli F, Kaiser C, Iglesias JF, Jan van Geuns R, Daemen J, Spirk D, Engstrom T, Lang I, Windecker S, Koskinas KC, Losdat S, Raber L. Impact of alirocumab on plaque regression and haemodynamics of non-culprit arteries in patients with acute myocardial infarction: a prespecified substudy of the PACMAN-AMI trial. EuroIntervention. 2023 Jul 17;19(4):e286-e296. doi: 10.4244/EIJ-D-23-00201. PMID 37341586
- [Derived] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058
- [Derived] Zanchin C, Koskinas KC, Ueki Y, Losdat S, Haner JD, Bar S, Otsuka T, Inderkum A, Jensen MRJ, Lonborg J, Fahrni G, Ondracek AS, Daemen J, van Geuns RJ, Iglesias JF, Matter CM, Spirk D, Juni P, Mach F, Heg D, Engstrom T, Lang I, Windecker S, Raber L. Effects of the PCSK9 antibody alirocumab on coronary atherosclerosis in patients with acute myocardial infarction: a serial, multivessel, intravascular ultrasound, near-infrared spectroscopy and optical coherence tomography imaging study-Rationale and design of the PACMAN-AMI trial. Am Heart J. 2021 Aug;238:33-44. doi: 10.1016/j.ahj.2021.04.006. Epub 2021 May 2. PMID 33951415